CLINICAL TRIAL: NCT01065714
Title: Transepidermal Water Loss (TEWL) and Corneometry With Hydrogel Vehicle in the Treatment of Atopic Dermatitis - A Randomized, Investigator-Blind Pilot Study
Brief Title: A Study to Investigate the Use of Hydrogel Vehicle in Maintaining the Skin Barrier in Persons With Atopic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Derm Research, PLLC (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Leon Kircik, M.D., Principal Investigator, Derm Research, PLLC
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HGV0901
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Results first posted 2013-04-25 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2013-04

CONDITIONS: Atopic Dermatitis
Keywords: Transepidermal water loss; Epidermal barrier; Skin hydration
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Hydrogels

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydrogel vehicle (Experimental): Parallel designed study. Split body treatment
  Interventions: Drug: Hydrogel vehicle
- Eucerin Lotion (Active Comparator): Parallel study design. Split body study.
  Interventions: Drug: Eucerin Lotion

INTERVENTIONS:
Drug: Hydrogel vehicle — Each morning and evening, gently wash the target area with warm water and gently pat dry with soft towel. Once dry place a small amount of Hydrogel vehicle onto the tip of your finger. Place a dab of the Hydrogel vehicle on either the left or right side of the body as instructed. (Do not use Hydrogel vehicle and Eucerin lotion on the same side of the body.)
  Arms: Hydrogel vehicle
Drug: Eucerin Lotion — Each morning and evening, gently wash the area with warm water and pat dry with a soft towel. Once dry, place a small amount of Eucerin lotion to the target area on either the left or right side of the body as instructed. (Do not use Eucerin and Hydrogel vehicle on the same side of the body.)
  Arms: Eucerin Lotion

SUMMARY:
While the repair of the epidermal barrier in atopic dermatitis is of major importance in the treatment of atopic dermatitis, most of the vehicles used may actually cause a worsening of an impaired epidermal barrier. Hydrogel vehicle is anecdotally known to be moisturizing and hydrating.This study will compare the use of Hydrogel vehicle and Eucerin Lotion in maintaining the epidermal barrier in subjects with atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Definitive diagnosis of atopic dermatitis as characterized by Hanifin and Rajka criteria:
* 3 out of 4 major characteristics
* At least 3 minor characteristics
* Mild to moderate disease score of 2 or 3 by Investigator Global Assessment
* Minimum 5% Body Surface Area at Baseline
* Uniformly bilateral signs and symptoms of atopic dermatitis
* Able to understand and comply with the requirements of the study and sign Informed Consent/HIPAA forms. Subjects under the legal age of consent must also have written informed consent of the parent or legal guardian.

Exclusion Criteria:

* Allergy or sensitivity to any component of the test articles.
* Subjects who have not complied with the proper washout periods for prohibited medications.
* Significant coagulation disorder or any medical condition that, in the opinion of the investigator, contraindicates the subject's participation in the study.
* Recent alcohol or drug abuse is evident.
* History of poor cooperation, non-compliance with medical treatment or unreliability
* Participation in an investigational drug study within 30 days of the Baseline Visit.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-02; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leon H. Kirick, M.D., Principal Investigator — DermResearch, PLLC
Locations (1):
- DermResearch, PLLC, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from March 2010 through September 2010. Subjects enrolled from physician data base.
Groups:
- Hydrogel Vehicle/Eucerin Lotion: Parallel designed study. Split body treatment. Eucerin Lotion applied to one side of body, Hydrogel applied to the opposite side of body.
Period: Overall Study
Arm/Group | Hydrogel Vehicle/Eucerin Lotion
Started | 20 (This was a "split body" Study. All participants used both Hydrogel and Eucerin)
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Hydrogel Vehicle/Eucerin Lotion: Parallel designed study. Split body treatment
Arm/Group | Hydrogel Vehicle/Eucerin Lotion
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 15
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 35 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Percent Change of Trans Epidermal Water Loss (TEWL) With Use of Eucerin Lotion
Description: The average of three sequential Tewameter 300 meter readings taken at a minimum of one minute intervals on targeted area of body half treated with Eucerin lotion
Time Frame: Day 1 to Day 14
Population: per protocol
Measure: Median (Full Range); unit: percent change
Groups:
- Skin Barrier Function With Eucerin Lotion: Measurement of TEWL on targeted area on one side of body treated with Eucerin Lotion
Arm/Group | Skin Barrier Function With Eucerin Lotion
Number analyzed (Participants) | 20
percent change | 21.4 (54.8) [-66.8 to 214.8]

2. Primary Outcome: Percent Change of Trans Epidural Water Loss (TEWL) With the Use of Hydrogel Vehicle
Description: The average of three sequential Tewameter 300 meter readings taken at a minimum of one minute intervals on target areas of body half treated with Hydrogel vehicle
Time Frame: Day 1 to Day 14
Population: Per protocol
Measure: Median (Full Range); unit: percent change
Groups:
- Skin Barrier Function With Hydrogel Vehicle: Trans epidural water loss measurements on target areas of body side treated with Hydrogel vehicle
Arm/Group | Skin Barrier Function With Hydrogel Vehicle
Number analyzed (Participants) | 20
percent change | 4.2 (31.2) [-76.9 to 57.9]

3. Secondary Outcome: Percentage of Participants With an Increase in Skin Hydration Using Eucerin Lotion on Targeted Area on One Half of Body
Description: Five timed readings ( 0, 15, 30, 45 and 60 minutes) were taken using the Corneometer 825 meter on subjects using Eucerin lotion on targeted area on one half of body
Time Frame: Baseline to 14 days
Population: per protocol
Measure: Mean (Standard Deviation); unit: Percentage of participants
Groups:
- Skin Hydration With Eucerin: Parallel designed study. Split body treatment. Five corneometer readings were taken on the targeted area of one half of the body on which Eucerin Lotion was applied.
Arm/Group | Skin Hydration With Eucerin
Number analyzed (Participants) | 20
Percentage of participants | 33.5 (72.2)

4. Secondary Outcome: Percentage of Participants With an Increase in Skin Hydration Using Hydrogel Vehicle on Targeted Area of One Half of Body.
Description: Five timed readings at (0, 15, 30, 45 and 60 minutes) were taken, using the Corneometer 825 meter, on participants using Hydrogel vehicle
Time Frame: Baseline to 14 days
Population: per protocol
Measure: Mean (Standard Deviation); unit: percentage of participants
Groups:
- Skin Hydration With Hydrogel: Parallel designed study. Split body treatment. Hydrogel vehicle applied to targeted area one side of body. Skin Hydration measured by 5 Corneometer readings.
Arm/Group | Skin Hydration With Hydrogel
Number analyzed (Participants) | 20
percentage of participants | 32.3 (51.5)

ADVERSE EVENTS:
Arm/Group | Hydrogel Vehicle/Eucerin Lotion
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
Small number of participants, pilot study, short term

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes